CLINICAL TRIAL: NCT01272804
Title: A Phase 1 Placebo-controlled Trial To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Multiple Escalating Oral Doses Of Pf-04937319 In Adult Patients With Type 2 Diabetes Mellitus (t2dm)
Brief Title: Multiple Dose Study Of PF-04937319 In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1621003
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2; NIDDM
Keywords: Pharmacokinetics PK Pharmacodynamics PD T2DM Phase 1 Type 2 diabetes mellitus safety and tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N,N-dimethyl-5-((2-methyl-6-((5-methylpyrazin-2-yl)carbamoyl)benzofuran-4-yl)oxy)pyrimidine-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04937319 (Experimental)
  Interventions: Drug: PF-04937319
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04937319 — Subjects will be dosed with PF-04937319 for 14 days. The doses planned are 10, 30, 100 and 300 mg QD. All doses will be administered as tablets (10 and 100 mg strengths). In each Cohort, 9 patients will receive PF 04937319 and 3 will receive placebo. An additional cohort of 12 patients (9 active, 3 placebo) may be performed to explore a QD or BID dose. The dose for this additional cohort could be a dose already studied or a new dose that is within the exposure stopping criteria.
  Arms: PF-04937319
Drug: Placebo — Placebo to match PF-04937319 will be provided. Subjects will be dosed for 14 days. In each cohort 9 subjects will receive PF-04937319 and 3 will receive placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of PF-04937319 following multiple (14 days) escalating oral doses in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who are taking metformin only.
* Treatment should be stable, where this is defined as no change in the treatment, including dose, over the past 2 months. Regimens may include once daily and twice daily dosing only.
* Male and/or female patients (females will be women of non childbearing potential)
* Body Mass Index (BMI) of 18.5 to 45.0 kg/m2; and a total body weight >50 kg (110 lbs).
* HbA1c between 7.0% and 10.0%.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). Patients who have chronic conditions other than T2DM (for example, hypercholesterolemia or hypertension) but are controlled by either diet or stable (for the last 2 months) doses of medications may be included as well (for example, a subject with hypercholesterolemia on appropriate treatment is eligible).
* Evidence or history of diabetic complications with significant end organ damage, eg, proliferative retinopathy and/or macular edema, creatinine clearance less than 60 mL/min
* Any condition possibly affecting drug absorption (eg, gastrectomy)
* History of stroke or transient ischemic attack or myocardial infarction within the past 6 months
* History of coronary artery bypass graft or stent implantation.
* Clinically significant peripheral vascular disease (eg, manifested by claudication).
* Any history or clinical evidence of congestive heart failure, NYHA Classes II to IV.
* One or more self reported significant/severe/requiring treatment episodes of hypoglycemia within the last 3 months, or two or more self reported significant/severe/requiring treatment episodes of hypoglycaemia within the last 6 months.
* Current history of angina/unstable angina.
* Milk or soy allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Elite Research Institute, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio

REFERENCES:
- [Derived] Sharma R, Litchfield J, Atkinson K, Eng H, Amin NB, Denney WS, Pettersen JC, Goosen TC, Di L, Lee E, Pfefferkorn JA, Dalvie DK, Kalgutkar AS. Metabolites in safety testing assessment in early clinical development: a case study with a glucokinase activator. Drug Metab Dispos. 2014 Nov;42(11):1926-39. doi: 10.1124/dmd.114.060087. Epub 2014 Aug 20. PMID 25142735
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621003&StudyName=Multiple%20Dose%20Study%20Of%20PF-04937319%20In%20Patients%20With%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04937319 10 mg: Participants received PF-04937319 10 milligram (mg) tablet orally once daily for 14 days.
- PF-04937319 30 mg: Participants received PF-04937319 30 mg (3 tablets of 10 mg) orally once daily for 14 days.
- PF-04937319 50 mg: Participants received PF-04937319 50 mg (5 tablets of 10 mg) orally once daily for 14 days.
- PF-04937319 100 mg: Participants received PF-04937319 100 mg tablet orally once daily for 14 days.
- PF-04937319 300 mg: Participants received PF-04937319 300 mg (3 tablets of 100 mg) orally once daily for 14 days.
- Placebo: Participants received placebo matched to PF-04937319 tablet orally once daily for 14 days.
Period: Overall Study
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Started | 9 | 9 | 9 | 9 | 9 | 16
Completed | 8 | 9 | 9 | 9 | 7 | 15
Not Completed | 1 | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.2) | 49.4 (7.8) | 54.2 (5.4) | 51.4 (10.6) | 56.4 (5.8) | 57.3 (5.8) | 54.4 (7.7)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 0 | 2 | 3 | 3 | 6 | 18
  Male | 5 | 9 | 7 | 6 | 6 | 10 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 14 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline (Day 1) up to 14 days after last dose of study treatment (up to 28 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
participants
  AEs | 6 | 5 | 0 | 3 | 8 | 5
  SAEs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) On Day 1
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours (hrs) post morning dose on Day 1 (fasted condition)
Population: Pharmacokinetic (PK) parameter analysis population included all enrolled participants treated with PF-04937319 who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
nanogram per milliliter (ng/mL) | 38.22 (25) | 69.49 (32) | 119.4 (38) | 245.4 (42) | 449.3 (39)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) On Day 6
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8 hours post-dose on Day 6 (fed condition)
Population: PK parameter analysis population included all enrolled participants treated with PF-04937319 who had at least 1 of the PK parameters of interest. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 7
ng/mL | 57.73 (17) | 122.3 (17) | 234.1 (24) | 421.5 (31) | 970.6 (35)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 1
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 1 (fasted condition)
Population: PK parameter analysis population included all enrolled participants treated with PF-04937319 who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
hour | 3.00 [1.50 to 8.00] | 3.00 [1.50 to 8.00] | 3.00 [2.95 to 5.00] | 3.00 [3.00 to 5.00] | 3.00 [1.50 to 8.00]

5. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 6
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8 hours post-dose on Day 6 (fed condition)
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 7
hour | 1.50 [1.50 to 5.05] | 1.50 [1.50 to 5.00] | 1.50 [1.50 to 8.00] | 1.50 [1.50 to 5.00] | 1.50 [0.50 to 5.07]

6. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) on Day 1
Description: AUCtau is the area under the plasma concentration versus time curve from time zero (pre-dose) to the end of the dosing interval (tau), here dosing interval is 24 hours.
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 1 (fasted condition)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
nanogram*hour per milliliter | 407.0 (29) | 867.7 (21) | 1456 (48) | 2749 (38) | 6034 (40)

7. Primary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax, ss) On Day 14
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 14 (fasted condition)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
ng/mL | 51.09 (27) | 79.30 (31) | 171.3 (36) | 251.5 (44) | 555.9 (44)

8. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration at Steady State (Tmax, ss) on Day 14
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 14 (fasted condition)
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
hour | 3.00 [1.50 to 3.02] | 3.00 [1.50 to 8.00] | 3.00 [3.00 to 8.00] | 3.00 [3.00 to 8.00] | 3.00 [3.00 to 8.00]

9. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval at Steady State (AUCtau, ss) on Day 14
Description: AUCtau, ss = Area under the plasma concentration versus time curve from time zero (pre-dose) to the end of the dosing interval (tau) at steady state, here dosing interval is 24 hours.
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 14 (fasted condition)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
nanogram*hour per milliliter | 458.0 (35) | 928.7 (23) | 1889 (52) | 3167 (40) | 7446 (42)

10. Primary Outcome: Plasma Decay Half-Life (t1/2) on Day 14
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24, 36, 48 hours post morning dose on Day 14 (fasted condition)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
hour | 6.563 (0.77897) | 6.884 (1.9264) | 6.348 (1.4271) | 6.960 (1.0358) | 8.479 (2.4173)

11. Primary Outcome: Minimum Observed Plasma Trough Concentration at Steady State (Cmin, ss) on Day 14
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16 hours post morning dose on Day 14 (fasted condition)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
ng/mL | 1.380 (83) | 10.56 (43) | 22.73 (103) | 41.68 (64) | 129.8 (62)

12. Primary Outcome: Percentage of Unchanged Drug Excreted in the Urine Over Dosing Interval (Ae[%]) on Day 14
Description: Percentage of drug excreted unchanged in urine calculated as overall amount of unchanged drug excreted in the urine over the dosing interval (24 hours) divided by total daily dose multiplied by 100.
Time Frame: 0 hour (pre-dose) through 24 hours post-dose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 7 | 9 | 9 | 9 | 5
percentage of dose | 0.3904 (0.11901) | 0.3533 (0.20183) | 0.6463 (0.56717) | 0.5380 (0.34593) | 0.4294 (0.44676)

13. Primary Outcome: Apparent Oral Clearance (CL/F) on Day 14
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 14 (fasted condition)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
liter per hour | 21.86 (25) | 32.32 (23) | 26.48 (34) | 31.56 (37) | 40.29 (43)

14. Primary Outcome: Apparent Volume of Distribution (Vz/F) on Day 14
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 14 (fasted condition)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
liter | 205.3 (20) | 311.6 (32) | 236.7 (27) | 314.0 (28) | 475.2 (48)

15. Primary Outcome: Observed Accumulation Ratio for AUCtau (Rac)
Description: Accumulation ratio for AUCtau (Rac) was calculated as area under the curve from time zero to end of dosing interval (AUCtau) on Day 14 divided by area under the curve from time zero to end of dosing interval (AUCtau) on Day 1. Dosing interval = 24 hours.
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 1 and Day 14 (fasted condition)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
ratio | 1.204 (22) | 1.069 (15) | 1.296 (24) | 1.152 (22) | 1.118 (40)

16. Primary Outcome: Observed Accumulation Ratio for Cmax (Rac, Cmax)
Description: Accumulation ratio for Cmax (Rac, Cmax) was calculated as maximum observed plasma concentration (Cmax) on Day 14 divided by maximum observed plasma concentration (Cmax) on Day 1.
Time Frame: 0 (pre-dose), 0.5, 1.5, 3, 5, 8, 12, 16, 24 hours post morning dose on Day 1 and Day 14 (fasted condition)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 7
ratio | 1.414 (41) | 1.141 (28) | 1.437 (17) | 1.026 (25) | 1.080 (40)

17. Primary Outcome: Percent Change From Baseline in Glucose Area Under the Curve From Time 2 to 6 Hours (AUC [2-6]) After a Mixed Meal Tolerance Test (MMTT) at Day 1
Description: Percent change from baseline in area under the plasma glucose concentration-time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC. Baseline value was the AUC (2-6) calculated on Day -1.
Time Frame: -46, -45.75, -45.5, -45, -44.5, -44, -43, -42 hrs pre-dose on Day -1; 2, 2.25, 2.5, 3, 3.5, 4, 5, 6 hrs post-dose on Day 1 (fasted condition)
Population: Pharmacodynamic (PD) analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 PD parameter.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
percent change | -0.46 (8.881) | -2.67 (6.670) | 6.41 (14.532) | -12.11 (14.225) | -12.29 (13.711) | -3.71 (10.848)

18. Primary Outcome: Percent Change From Baseline in Glucose Area Under the Curve From Time 2 to 6 Hours (AUC [2-6]) After a Mixed Meal Tolerance Test (MMTT) at Day 14
Description: as for outcome 17
Time Frame: -46, -45.75, -45.5, -45, -44.5, -44, -43, -42 hrs pre-dose on Day -1; 2, 2.25, 2.5, 3, 3.5, 4, 5, 6 hrs post-dose on Day 14 (fasted condition)
Population: PD analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 PD parameter. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 6 | 15
percent change | -11.94 (15.477) | -4.91 (16.601) | -4.11 (17.321) | -26.83 (21.054) | -11.37 (15.205) | -2.86 (12.103)

19. Secondary Outcome: Percent Change From Baseline in Insulin Area Under the Curve From Time 2 to 6 Hours (AUC [2-6]) After a Mixed Meal Tolerance Test (MMTT) at Day 1 and 14
Description: Percent change from baseline in area under the plasma insulin concentration-time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC. Baseline value was the AUC (2-6) calculated on Day -1.
Time Frame: -46, -45.75, -45.5, -45, -44.5, -44, -43, -42 hrs pre-dose on Day -1; 2, 2.25, 2.5, 3, 3.5, 4, 5, 6 hrs post-dose on Day 1 and 14 (fasted condition)
Population: PD analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 PD parameter. Here 'n' signifies participants evaluable for this measure at specified time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
percent change
  Percent Change at Day 1 (n=9,9,9,9,9,16) | -2.22 (17.843) | 13.24 (22.221) | 24.11 (13.772) | 4.41 (17.470) | 18.10 (17.059) | -2.92 (15.768)
  Percent Change at Day 14 (n=8,9,9,9,7,15) | 15.77 (21.452) | 17.98 (26.499) | 30.86 (41.063) | 0.38 (21.140) | 39.23 (26.876) | 7.62 (26.034)

20. Secondary Outcome: Percent Change From Baseline in C-peptide Area Under the Curve From Time 2 to 6 Hours (AUC [2-6]) After a Mixed Meal Tolerance Test (MMTT) at Day 1 and 14
Description: Percent change from baseline in area under the plasma C-peptide concentration-time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC. Baseline value was the AUC (2-6) calculated on Day -1.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
percent change
  Percent Change at Day 1 (n=9,9,9,9,9,16) | -2.36 (10.170) | 8.53 (13.383) | 12.65 (9.974) | 2.37 (12.421) | 16.34 (8.940) | -1.43 (9.488)
  Percent Change at Day 14 (n=8,9,9,9,7,15) | 8.66 (11.069) | 13.49 (14.403) | 16.51 (27.962) | -1.44 (14.463) | 22.50 (14.809) | 1.80 (16.722)

21. Secondary Outcome: Change From Baseline in Average Plasma Glucose at Day 1, 6, 14
Description: Glucometer testing performed by finger-stick at 8 time points per day to measure glucose levels. Average plasma glucose was calculated as area under the plasma glucose concentration-time curve from 0 to 24 hours (AUC [0-24]) divided by 24.
Time Frame: -46, -44, -42, -40, -38, -36, -30, -27 hrs pre-dose on Day -1; 2, 6, 8, 10, 12,18,21 hrs post-dose on Day 1, 6 and 14; additional 0 hr (pre-dose) on Day 6 and 4 hr post-dose on Day 1 and 14
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
mg/dL
  Baseline (n=9,9,9,9,9,16) | 192.10 (22.913) | 188.83 (48.992) | 195.78 (37.871) | 205.38 (44.632) | 170.95 (51.465) | 189.07 (39.131)
  Change at Day 1 (n=9,9,9,9,9,16) | -7.18 (9.851) | -5.24 (6.421) | 8.72 (15.071) | -1.90 (21.784) | -23.26 (19.189) | 3.04 (17.611)
  Change at Day 6 (n=8,9,9,9,7,15) | -19.62 (16.247) | -6.35 (22.496) | 9.80 (30.359) | -32.36 (24.121) | -47.19 (25.752) | 3.92 (17.068)
  Change at Day 14 (n=8,9,9,9,7,15) | -12.65 (25.918) | -16.45 (27.709) | -14.79 (33.687) | -48.87 (27.216) | -34.15 (24.596) | -7.48 (21.703)

22. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Time Frame: Baseline (Pre-dose on Day 1), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
mg/dL
  Baseline (n=9,9,9,9,9,16) | 173.78 (31.952) | 181.33 (50.621) | 190.11 (34.505) | 193.67 (45.695) | 162.33 (50.269) | 172.44 (42.527)
  Change at Day 2 (n=9,9,9,9,9,16) | -5.00 (10.840) | -4.67 (12.845) | -6.78 (25.430) | -1.78 (14.507) | -23.44 (18.662) | 0.94 (12.588)
  Change at Day 3 (n=9,9,9,9,9,16) | -19.11 (10.216) | -5.78 (10.171) | -18.78 (27.124) | -13.22 (15.571) | -32.78 (17.527) | -7.81 (16.885)
  Change at Day 4 (n=9,9,9,9,8,16) | -13.44 (19.603) | -9.44 (16.001) | -13.78 (28.900) | -19.67 (20.899) | -42.88 (20.972) | -4.13 (18.722)
  Change at Day 5 (n=9,9,9,9,9,16) | -19.67 (16.256) | -9.89 (15.358) | -22.56 (29.560) | -26.56 (21.030) | -30.33 (22.170) | -14.06 (21.402)
  Change at Day 6 (n=9,9,9,9,7,15) | -10.89 (18.210) | -16.33 (17.804) | -18.00 (34.380) | -29.11 (16.027) | -43.00 (15.610) | -8.27 (12.708)
  Change at Day 7 (n=8,9,9,9,7,15) | -13.50 (21.314) | -12.78 (13.664) | -14.44 (37.270) | -30.22 (16.672) | -43.71 (18.117) | -5.60 (12.704)
  Change at Day 8 (n=8,9,9,9,7,15) | -23.25 (21.212) | -8.56 (20.415) | -5.56 (37.964) | -24.11 (19.934) | -31.71 (20.155) | -4.93 (16.434)
  Change at Day 9 (n=8,9,9,9,7,15) | -19.63 (20.784) | -22.11 (20.709) | -9.78 (42.825) | -24.78 (17.817) | -38.00 (19.502) | -2.80 (15.857)
  Change at Day 10 (n=8,9,9,9,7,15) | -23.88 (23.503) | -16.89 (20.847) | -16.33 (32.427) | -37.11 (19.877) | -34.29 (24.452) | -6.20 (10.544)
  Change at Day 11 (n=8,9,9,9,7,15) | -17.38 (28.540) | -22.56 (22.490) | -18.11 (39.810) | -32.89 (20.294) | -38.57 (22.240) | -5.73 (19.374)
  Change at Day 12 (n=8,9,9,9,7,15) | -27.13 (28.423) | -18.56 (28.183) | -16.89 (41.870) | -32.22 (17.880) | -43.57 (26.576) | -7.73 (17.910)
  Change at Day 13 (n=8,9,9,9,7,15) | -18.13 (30.258) | -23.44 (23.807) | -24.78 (40.822) | -30.89 (19.548) | -39.71 (22.706) | -12.27 (18.718)
  Change at Day 14 (n=8,9,9,9,7,15) | -33.63 (26.175) | -23.67 (25.441) | -26.56 (39.768) | -43.78 (22.725) | -41.86 (22.386) | -11.80 (16.545)
  Change at Day 15 (n=8,9,9,9,7,15) | -13.38 (22.595) | -21.44 (26.034) | -23.89 (38.238) | -44.11 (19.586) | -40.57 (25.553) | -11.47 (17.916)

23. Secondary Outcome: Change From Baseline in Triglyceride (TG) Level at Day 3, 6, 10, 14, 16 and Follow-up
Description: Blood sample for lipid biomarker was taken following 12-hours fasting. Baseline value was collected on Day -2 for lipids.
Time Frame: Baseline (Day -2), Day 3, 6, 10, 14, 16 and Follow-up (7 to 14 days after last dose of study medication)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
mg/dL
  Baseline (n=9,9,9,9,9,16) | 178.89 (63.21) | 152.33 (43.88) | 175.56 (53.32) | 192.78 (91.62) | 123.33 (47.89) | 152.31 (70.46)
  Change at Day 3 (n=9,9,9,9,9,16) | -5.89 (82.19) | 1.67 (63.16) | -44.44 (45.88) | -25.44 (59.99) | 0.22 (42.40) | 0.88 (47.31)
  Change at Day 6 (n=9,9,9,9,7,15) | -32.00 (70.40) | -1.33 (65.02) | -40.44 (50.85) | -29.00 (62.90) | 13.14 (51.50) | -14.67 (51.85)
  Change at Day 10 (n=8,9,9,9,7,15) | -16.88 (58.15) | 1.78 (66.28) | -6.44 (59.39) | -13.56 (51.83) | 30.71 (43.77) | 2.13 (46.04)
  Change at Day 14 (n=8,9,9,9,7,15) | -19.25 (76.20) | -4.44 (65.79) | -37.33 (48.75) | -40.33 (55.72) | 15.57 (38.25) | -21.67 (44.03)
  Change at Day 16 (n=8,9,9,9,7,14) | 13.25 (108.99) | -6.67 (80.27) | -36.22 (50.27) | -35.33 (53.61) | 23.57 (50.04) | -19.07 (47.96)
  Change at Follow-up (n=9,9,9,9,7,16) | -41.22 (73.73) | 38.78 (163.30) | 4.56 (73.52) | -45.44 (120.43) | 22.29 (57.79) | 1.94 (52.43)

24. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) Level at Day 3, 6, 10, 14, 16 and Follow-up
Description: as for outcome 23
Time Frame: Baseline (Day -2), Day 3, 6, 10, 14, 16 and Follow-up (7 to 14 days after last dose of study medication)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
mg/dL
  Baseline (n=9,9,9,9,9,16) | 200.56 (34.32) | 207.33 (41.11) | 205.00 (50.52) | 213.22 (53.38) | 170.22 (41.37) | 181.94 (34.45)
  Change at Day 3 (n=9,9,9,9,9,16) | -24.00 (17.21) | -9.33 (13.46) | -14.22 (16.93) | -16.33 (18.33) | -11.56 (31.13) | -7.50 (18.40)
  Change at Day 6 (n=9,9,9,9,7,15) | -19.11 (20.95) | -25.11 (19.47) | -20.78 (19.39) | -11.33 (21.17) | 0.00 (42.90) | -6.47 (26.19)
  Change at Day 10 (n=8,9,9,9,7,15) | -30.00 (24.51) | -14.67 (14.40) | -30.89 (17.41) | -15.11 (20.76) | -2.29 (41.43) | 0.33 (30.00)
  Change at Day 14 (n=8,9,9,9,7,15) | -31.50 (21.08) | -29.11 (14.42) | -27.44 (17.08) | -24.22 (25.73) | 1.29 (41.63) | -6.60 (37.37)
  Change at Day 16 (n=8,9,9,9,7,14) | -26.38 (26.72) | -22.11 (13.60) | -29.11 (20.26) | -12.11 (24.49) | 1.86 (45.05) | -1.43 (32.90)
  Change at Follow-up (n=9,9,9,9,7,16) | -19.44 (25.73) | -12.44 (24.70) | -29.44 (27.13) | -33.56 (40.73) | -15.29 (8.24) | -5.50 (29.57)

25. Secondary Outcome: Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C) Level at Day 3, 6, 10, 14, 16 and Follow-up
Description: as for outcome 23
Time Frame: Baseline (Day -2), Day 3, 6, 10, 14, 16 and Follow-up (7 to 14 days after last dose of study medication)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
mg/dL
  Baseline (n=9,9,9,9,9,16) | 116.67 (37.41) | 133.56 (43.47) | 123.44 (35.72) | 130.67 (33.83) | 96.11 (37.88) | 102.44 (31.64)
  Change at Day 3 (n=9,9,9,9,9,16) | -19.22 (22.22) | -5.89 (19.37) | -6.89 (15.26) | -6.67 (19.46) | -11.00 (23.51) | -3.63 (14.80)
  Change at Day 6 (n=9,9,9,9,7,15) | -8.78 (23.21) | -20.44 (22.32) | -13.67 (14.74) | -2.33 (22.11) | -0.29 (38.98) | 2.73 (20.35)
  Change at Day 10 (n=8,9,9,9,7,15) | -19.00 (24.94) | -11.44 (16.84) | -30.89 (14.08) | -7.89 (17.92) | -9.57 (35.69) | 5.07 (24.99)
  Change at Day 14 (n=8,9,9,9,7,15) | -17.13 (21.14) | -22.44 (16.49) | -19.89 (14.68) | -11.56 (17.92) | -1.00 (38.18) | 4.80 (30.59)
  Change at Day 16 (n=8,9,9,9,7,14) | -17.88 (22.22) | -15.00 (14.11) | -20.22 (16.75) | -0.67 (16.86) | -3.86 (38.21) | 5.79 (27.50)
  Change at Follow-up (n=9,8,9,9,7,16) | -6.22 (24.40) | -10.38 (15.15) | -27.11 (22.05) | -19.78 (22.97) | -17.43 (16.70) | -2.25 (23.61)

26. Secondary Outcome: Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C) Level at Day 3, 6, 10, 14, 16 and Follow-up
Description: as for outcome 23
Time Frame: Baseline (Day -2), Day 3, 6, 10, 14, 16 and Follow-up (7 to 14 days after last dose of study medication)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
mg/dL
  Baseline (n=9,9,9,9,9,16) | 48.11 (10.96) | 43.33 (9.51) | 46.44 (11.51) | 43.89 (13.66) | 49.44 (14.05) | 48.94 (9.33)
  Change at Day 3 (n=9,9,9,9,9,16) | -3.56 (4.10) | -3.67 (6.36) | 1.33 (6.75) | -4.56 (4.07) | -0.67 (7.07) | -3.88 (8.02)
  Change at Day 6 (n=9,9,9,9,7,15) | -4.00 (2.65) | -4.33 (7.73) | 1.00 (4.66) | -3.11 (3.69) | -2.43 (2.64) | -6.20 (7.80)
  Change at Day 10 (n=8,9,9,9,7,15) | -7.63 (4.21) | -3.44 (5.98) | 1.22 (5.70) | -4.44 (3.21) | 1.14 (4.49) | -5.00 (7.99)
  Change at Day 14 (n=8,9,9,9,7,15) | -10.50 (5.78) | -5.78 (10.59) | 0.00 (5.15) | -4.44 (4.93) | -0.86 (4.38) | -6.93 (9.52)
  Change at Day 16 (n=8,9,9,9,7,14) | -11.0 (5.10) | -5.78 (7.61) | -1.56 (5.70) | -4.22 (4.12) | 1.00 (3.79) | -3.36 (9.04)
  Change at Follow-up (n=9,9,9,9,7,16) | -4.89 (3.98) | -5.22 (6.50) | -3.22 (7.24) | -4.44 (6.98) | -2.29 (4.07) | -3.50 (6.86)

27. Secondary Outcome: Change From Baseline in Lactate Level at Day 6 and 14
Description: Baseline value was collected at 0 hour on Day 1 for lactate.
Time Frame: Baseline (Day 1), Day 6 and 14
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 16
mg/dL
  Baseline (n=9,9,9,9,9,16) | 17.64 (5.14) | 10.17 (3.07) | 14.14 (7.82) | 21.66 (9.45) | 11.57 (4.30) | 14.74 (8.58)
  Change at Day 6 (n=9,9,9,9,7,15) | -2.44 (7.95) | 1.02 (1.77) | -2.08 (7.14) | -6.08 (10.72) | 2.61 (6.60) | -1.45 (9.27)
  Change at Day 14 (n=8,9,9,9,7,15) | 0.21 (3.07) | -0.09 (2.02) | -3.88 (6.63) | -6.97 (10.42) | 2.60 (2.98) | -2.59 (8.67)

ADVERSE EVENTS:
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 50 mg | PF-04937319 100 mg | PF-04937319 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/16
Other Adverse Events (participants affected / at risk) | 6/9 | 5/9 | 0/9 | 3/9 | 8/9 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04937319 10 mg (N=9) | PF-04937319 30 mg (N=9) | PF-04937319 50 mg (N=9) | PF-04937319 100 mg (N=9) | PF-04937319 300 mg (N=9) | Placebo (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 6 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.